CLINICAL TRIAL: NCT00161681
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Levonorgestrel 90 Mcg and Ethinyl Estradiol 20 Mcg in a Continuous Daily Regimen on Menstrual Cycle-Related Symptoms
Brief Title: Study Evaluating Levonorgestrel/Ethinyl Estradiol (LNG/EE) in PMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0858A2-322; B3121024 (Other: Pfizer)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2007-05

CONDITIONS: Premenstrual Syndrome
Keywords: Levonorgestrel; ethinyl estradiol; premenstrual syndrome; menstrual cycle related symptoms
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Ethinyl Estradiol-Norgestrel Combination

INTERVENTIONS:
Drug: Levonorgestrel/Ethinyl Estradiol

SUMMARY:
The purpose of this study is to determine whether LNG/EE is effective in the treatment of menstrual cycle related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18 to 49 years
* Regular 21 to 35 day menstrual cycles for 3 months prior to study visit 1
* History of menstrual cycle related symptoms as determined by the investigator.

Exclusion Criteria:

* Contraindication to combination oral contraceptives
* Depression requiring hospitalization or associated with suicidal ideation within the last 3 years
* Use of antidepressants/anxiolytics within 10 days of screening and for the duration of the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 2005-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of a continuous-use OC regimen containing a combination of LNG/EE in preventing moderate to severe cycle-related symptoms compared with placebo

SECONDARY OUTCOMES:
To evaluate the effects of this LNG/EE regimen on work productivity and subject satisfaction in subjects with moderate to severe cycle-related symptoms at baseline compared with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (43):
- United States (43):
  - Huntsville, Alabama
  - Peoria, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - San Diego, California
  - Denver, Colorado
  - Longmont, Colorado
  - Aventura, Florida
  - Boynton Beach, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Fort Myers, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Lexington, Kentucky
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Moorestown, New Jersey
  - Rochester, New York
  - Fayetteville, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Mogadore, Ohio
  - Eugene, Oregon
  - Medford, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wexford, Pennsylvania
  - Hilton Head Island, South Carolina
  - Mt. Pleasant, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Sandy City, Utah
  - Richmond, Virginia
  - Lakewood, Washington
  - Seattle, Washington